CLINICAL TRIAL: NCT03853603
Title: Clinical Study to Investigate the Effects of a Food Supplement With Santa Herba Extract on Weight Loss and Modulation of Appetite-related Biomarkers in Overweight Women - a Randomized, Placebo-controlled Parallel Study
Brief Title: Clinical Study to Investigate the Effects of a Food Supplement Santa Herba Extract on Weight Loss in Overweight Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mibelle AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BTS1235/18
Record Dates: First submitted 2019-02-12; First posted 2019-02-25 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Weight Loss
Keywords: lipid profile; 12,13-diHOME
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Placebo
- Santa herba extract (Active Comparator): Santa herba extract
  Interventions: Dietary Supplement: Santa herba

INTERVENTIONS:
Dietary Supplement: Santa herba — Santa herba dry extract; 400 mg/day. 2 capsules/day; 1 capsule twice daily with the main meals (lunch and dinner)
  Arms: Santa herba extract
Dietary Supplement: Placebo — Maltodextrin; 400 mg/day. 2 capsules/day; 1 capsule twice daily with the main meals (lunch and dinner)
  Arms: Placebo

SUMMARY:
Aim of the study is to investigate the effect of a 12-week supplementation of Santa Herba Extract on body weight in overweight and obese subjects. Additionally appetite related marker as well as marker of white adipose tissue browning will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able and willing to follow the study protocol procedures to sign the Informed Consent Form prior to screening evaluations
* Overweight and obese women with BMI 25 - 35 kg/m2 (limits included)
* Age: 25 - 60 years
* Subject is in good physical and mental health as established by medical history, physical examination, electrocardiogram, vital signs, results of biochemistry, haematology

Exclusion Criteria:

* Relevant history or presence of any medical disorder potentially interfering with this study (heavy depression, diabetes, active cancer, severe liver disease, heavy cardiovascular diseases (e.g. stroke, heart attack))
* Chronic intake of medication/dietary supplements with impact on body weight or body composition or lipid modifying products (e.g. protein shakes, statins, omega-3 fatty acids, etc.) 2 months prior to screening or during the study; stable doses of e.g. hypertensive therapy and thyroid gland hormones are acceptable.
* Change in hormonal contraceptive during or at least 3 months before the study
* Consumption of any dietary supplement / fortified food (with exception of vitamin D and mineral supplements e.g. Ca, Mg)
* Low body fat mass measured at screening with BIA ( bioelectrical impedance analysis ) (Cut off-value: <36% body fat).
* Weight loss intervention or recent body weight change > 4.5 kg during last 3 months
* Diet high in vegetables and fruits ≥ 5 portions per day
* Vegan lifestyle
* Smoker > 10 cigarettes / day
* Gastrointestinal diseases/conditions (colitis ulcerosa, Crohn's disease, peptic ulcers, celiac disease)

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
Body weight | day 85
  electronic scale

SECONDARY OUTCOMES:
Body fat (%) | Day 85
  Body fat mass in kilograms (kg) and weight in kilograms (kg) will be combined to report Percent body fat in (kg/kg)*100 (%)
BCM/ECM index | Day 85
  Body cell mass (BCM) in kg and extracellular mass (ECM) in kg will be combined to report BCM/ECM index
Waist-hip ratio (WHR) | Day 85
  Waist circumference in centimetre (cm) and hip circumference in centimetre (cm) will be combined to report WHR in cm/cm
Sagittal abdominal diameter (SAD) [cm] | Day 85
  Sagittal abdominal diameter (SAD) or "supine abdominal height" is a simple anthropometric measure shown to be a marker of insulin resistance. SAD is measured after normal expiration at the level of iliac crest while in the supine position with bent knees on a firm examination table and without clothes in the measurement area. The measurement is performed with the Holtain-Kahn abdominal caliper.
Concentration of lipid profile in serum | Day 85
  Concentration of Cholesterol [mg/dL], triglycerides [mg/dL], LDL-cholesterol [mg/dL], HDL-cholesterol [mg/dL]
Concentration of Lipokin in plasma | Day 85
  12,13-diHOME (12,13-Dihydroxyoctadec-9-enoic acid) [pmol/mL]
Questionnaire about Appetite (AEBQ) | Day 85
  The Adult Eating Behavior Questionnaire (Hunot et al. 2016) about perception of hunger and satiety including ravenousness appetite and snacking habits will be performed throughout the study. AEBQ is a questionnaire measuring 8 different appetitive traits.
  Enjoyment of food
  Emotional over-eating
  Emotional under-eating
  Food fussiness
  Food responsiveness
  Slowness in eating
  Hunger
  Satiety responsiveness
  Scale: 5-point Likert scale:
  Strongly disagree =1 Disagree =2 Neitheragree nor disagree =3 Agree =4 Strongly agree =5

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Menzel, MD, Principal Investigator — BioTeSys GmbH
Locations (1):
- BioTeSys GmbH, Esslingen am Neckar, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Modinger Y, Schon C, Wilhelm M, Pickel C, Grothe T. A Food Supplement with Antioxidative Santa Herba Extract Modulates Energy Metabolism and Contributes to Weight Management. J Med Food. 2021 Nov;24(11):1235-1242. doi: 10.1089/jmf.2021.0016. Epub 2021 Jul 13. PMID 34255555